CLINICAL TRIAL: NCT05513222
Title: Flipped Autograft: a Novel Approach for Management of Wound Dehiscence in Implant Dentistry
Brief Title: Flipped Autograft for Treating Surgical Wound Dehiscence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, assistant lecturer, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hamdy
Record Dates: First submitted 2022-08-20; First posted 2022-08-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flipped autograft (Experimental)
  Interventions: Procedure: flipped autograft

INTERVENTIONS:
Procedure: flipped autograft — Thick lingual flap was de-epithelized and partially dissected to increase its length then flipped and sutured to the buccal flap to obtain primary closure

SUMMARY:
This case report describes a novel technique for management of peri-implant wound dehiscence that involves using auto graft from the same surgical site to seal the dehiscence defect.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients in a healthy systemic condition.
2. Both genders
3. Patients should have single missing tooth.
4. Seibert Class I ridge defect.
5. Patients should approve to deliver a signature to a written consent after study nature explanation.

Exclusion Criteria:

* 1- Patients with any smoking habits. 2- Pregnant females, decisional impaired individuals, Prisoners and handicapped patients.

  3- Patients having poor oral hygiene or not wanting to carry out oral hygiene measures.

  4- Patients with infections either periodontally or periapically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
complete primary intention healing of the wound dehiscence | 3 months
  complete uneventful healing will be assessed clinically by measuring soft tissue width and thickness using periodontal probe under local anesthesia

SECONDARY OUTCOMES:
esthetic outcome and patient satisfaction. | 3 months
  esthetic outcome will be measured using pink esthetic score. Pink esthetic score (PES) will be recorded for five variables: "mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue color and texture at the facial aspect of the implant site". A score of 2, 1, or 0 will be assigned to all five parameters.
  also patient satisfaction will be recorded using:
  • (VAS) Visual analogue scale to measure postoperative pain. Pain score reported by the patient. directly through Visual Analogue Scale score (from 0 to 10. 0: no pain, 1: minimal pain, 5: moderate pain, 10: severe pain) which will be recorded after 2 weeks (Yildirim et al., 2017)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hamdy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided